CLINICAL TRIAL: NCT05954715
Title: Does Ischaemic Preconditioning Improve Upper Body Exercise Performance in People With Spinal Cord Injury? A Feasibility Study
Brief Title: Ischaemic Preconditioning and Upper Body Exercise Performance in Persons With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loughborough University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sven Hoekstra, Lecturer in Physiology and Rehabilitation Sciences, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STH22013
Record Dates: First submitted 2023-06-30; First posted 2023-07-20 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries
Keywords: Exercise capacity; Tolerability; Ischaemic preconditioning; Maximal voluntary contraction; Time to task failure; Fatigue
MeSH Terms: conditions — Spinal Cord Injuries; Fatigue | interventions — Ischemic Preconditioning; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Acute single blind randomised controlled trial
Who Masked: Participant
Masking Description: Both Sham and IPC consist of 5 min bouts of cuff inflation, using an identical cuff. While the applied pressure will differ between conditions, this will not be communicated with the study participants prior to the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC (Ischaemic Preconditioning) (Experimental): IPC will be administered to the upper limb using cuff inflation pressures of 200 mmHg or 60mm Hg above the systolic BP (whichever is higher). Four cycles of cuff inflation each lasting 5 min in duration followed by a 5-min period of cuff deflation will be applied.
  Interventions: Other: Ischaemic Preconditioning
- Sham (Sham Comparator): The Sham intervention will be administered with a BP cuff over the upper arm being inflated at a pressure 30mmg Hg below the diastolic blood pressure. The sham cycles will comprise of four cycles of cuff inflation each lasting 5 min in duration followed by a 5-min period of cuff deflation.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Ischaemic Preconditioning — Four cycles of cuff inflation each lasting 5 min in duration followed by a 5-min period of cuff deflation will be applied.
  Arms: IPC (Ischaemic Preconditioning)
Other: Sham — Four cycles of cuff inflation each lasting 5 min in duration followed by a 5-min period of cuff deflation will be applied.
  Arms: Sham

SUMMARY:
Regular physical activity improves physical fitness, fatigue, quality of life, gait and reduces progression of the disability in persons with SCI. However, persons with SCI are less physically active than the general population. Approximately 50% of people with SCI experience fatigue which impacts their daily activities.

Ischaemic preconditioning (IPC) is exposure of the body to brief periods of circulatory occlusion and reperfusion to protect organs against ischaemic injury. Recent studies have shown that IPC also improves exercise performance in healthy participants. The aim of this study is to determine whether it is feasible to use IPC to improve upper-body exercise performance in people with SCI.

Setting: Potential candidates will be identified from the Outpatient clinic at the Princess Royal Spinal Injuries Hospital (PRSCIC), Northern General Hospital, Sheffield.

Design: Acute single blind randomised controlled trial. Forty patients with SCI above 18 years and with preserved triceps function to conduct triceps strength testing will be randomised to receive either an IPC or sham intervention.

Interventions: IPC will be administered to the upper limb using cuff inflation pressures of 200 mmHg or 60mm Hg above the systolic BP (whichever is higher). Four cycles of cuff inflation each lasting 5 min in duration followed by 5-min period of cuff deflation will be applied. The Sham intervention will be administered with a BP cuff over the upper arm being inflated at a pressure 30mmg Hg below the diastolic blood pressure. The sham cycles will comprise of four cycles of cuff inflation each lasting 5 min in duration followed by 5-min period of cuff deflation.

Researchers will assess the feasibility of IPC as well as its efficacy to improve triceps maximal voluntary contraction and endurance compared with Sham.

DETAILED DESCRIPTION:
Once participants have signed informed consent, they will undergo the following procedures:

A. Randomisation into IPC vs Sham group B. Researcher will offer a suitable time to perform the study recording. C. Participant will be requested to spare up to 3 hours to complete the intervention.

D. Intervention session (IPC / Sham):

* Participant arrives.
* On arrival, after 10 minutes of seated rest, baseline heart rate and blood pressure (BP) will be measured.
* Two electrodes will be placed on the lateral triceps head for Electromyography (EMG) assessment during the triceps exercise capacity tests.
* To determine maximum voluntary contraction (MVC), a warm-up of 2 contractions each of a participant-estimated 50% MVC, 70% MVC, and 90% MVC, will first be performed. Participants will then undertake up to 5 maximal isometric contractions of the triceps, from which the MVC value will be obtained (average of the best 3 contractions).
* Following a rest period (5 minutes), a metronome will be used to give participants the cue to rhythmically isometrically contract their triceps (60 contraction-relaxation cycles/min) to a target value of 70% MVC.
* The time to task failure and ability to complete the exercise will be noted.
* Participants will report Rating of Perceived Exertion (RPE) using Borg's scale immediately after completing the exercise.
* Before and after the exercise, a capillary blood sample will be obtained from the earlobe for assessment of blood lactate concentration. Heart rate will be measured throughout.
* Repeat BP measurement.
* 30 minutes rest.
* Repeat BP and heart rate measurement.
* The MVC will be determined again, followed by a 5-minute rest.
* Proceed to intervention - 4 cycles of 5 minutes of IPC / Sham followed by 5 minutes of reperfusion. (Total 40 minutes).
* IPC intervention - This will involve tying the cuff of a manual BP apparatus around the upper arm and inflated to a minimum of 200 mmHg, or a pressure of 60 mmHg above the resting systolic BP, whichever is higher. The inflation will be maintained for 5 min followed by cuff deflation lasting 5 min. The cycle will be repeated four times.
* The Sham intervention will be delivered with the manual BP cuff tied to the upper arm. The cuff will be inflated 30 mm Hg below the diastolic BP for 5 min followed by deflation for 5 min. The cycle will be repeated four times.
* 10 minutes rest.
* Repeat pre-exercise capillary blood sample for determination of blood lactate concentration.
* Repeat 5 maximal isometric contractions of the triceps.
* Repeat a rest period of 5 min.
* Repeat rhythmic isometric triceps contraction exercise. Again, time to task failure and ability to complete the exercise will be noted.
* Repeat reading of Borg's Rating of Perceived Exertion (RPE) scale, post-exercise capillary blood sample, BP and heart rate measurements.
* Recording of adverse events and numerical pain scale, open ended discussion around perceptions and tolerability of IPC.
* 15 minutes rest.
* Repeat BP and heart rate measurement.
* Exit from study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older
* Chronic spinal cord injury (>1 year post injury)

Exclusion Criteria:

* ASIA Impairment scale E
* Other co-morbidities- Traumatic brain injury, Brachial plexus injury, upper limb fractures, progressive neurological conditions (e.g., multiple sclerosis)
* Patients known to have autonomic dysreflexia (AD) and having had an episode of AD in the last two weeks
* Impaired triceps function (medical research council (MRC) power motor score of 3 out of 5, or lower)
* Resting systolic BP of 170 mmHg or more
* Inability to communicate in English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | Recruitment figures and tolerability will be collected throughout the 1 year study period.
  The intervention will be considered feasible if all of the below criteria are met:
  * 80% of the target sample is recruited within the first 9 months after the start of recruitment.
  * Of those who participate, 80% tolerate the ischemic preconditioning intervention, defined as ratings <7 using the numerical Pain Rating Scale that ranges from 0 to 10. Here 0 is considered no pain; 1 to 3 is mild pain; 4 to 6 is moderate pain and 7 to 10 is severe pain.
  * A full data set is obtained in 80% of the participants who start the intervention.

SECONDARY OUTCOMES:
Maximal voluntary muscle contraction | Maximal voluntary muscle contraction will be collected throughout the 1 year study period.
  Maximal voluntary contraction of the triceps will be obtained before and after the intervention (IPC vs Sham).
Time to task failure during rhythmic muscle contraction | Time to task failure during rhythmic muscle contraction will be collected throughout the 1 year study period.
  Time to task failure during rhythmic triceps contraction will be obtained before and after the intervention (IPC vs Sham). The time that rhythmic triceps contractions at 70% of maximal voluntary contraction can be maintained will be recorded.

OTHER OUTCOMES:
Blood lactate concentration | Blood lactate concentration will be collected throughout the 1 year study period.
  Blood lactate concentration will be determined in a capillary blood sample obtained from the earlobe before and after the intervention.
Ratings of perceived exertion | Ratings of perceived extertion will be collected throughout the 1 year study period.
  Ratings of perceived exertion will be reported immediately following the exercise capacity tests of the triceps.
Electromyographic activity (EMG) at the triceps head | Electromyographic activity (EMG) at the triceps head will be collected throughout the 1 year study period.
  As an exploratory measure, EMG activity will be measured during the exercise capacity tests before and after the intervention at the head of the triceps. Fourier transformation of the EMG signal will be performed and compared between conditions at key time points as well as averaged over the entire test period.

CONTACTS AND LOCATIONS:
Overall Officials: Christof Leicht, PhD, Principal Investigator — Loughborough University

IPD SHARING:
Plan to Share IPD: No